CLINICAL TRIAL: NCT03808688
Title: A Multicenter, Open-label Study of Rhopressa® (Netarsudil Ophthalmic Solution) 0.02% for the Reduction of Elevated Intraocular Pressure in Patients With Glaucoma or Ocular Hypertension in a Real-world Setting
Brief Title: Study of Rhopressa® for the Reduction of Elevated Intraocular Pressure in Patients With Glaucoma or Ocular Hypertension in a Real-world Setting
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aerie Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-RHO-18-002
Record Dates: First submitted 2019-01-10; First posted 2019-01-17 (Actual); Results first posted 2020-09-29 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2019-11

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Netarsudil Ophthalmic Solution 0.02% (Other)
  Interventions: Drug: Netarsudil Ophthalmic Solution 0.02%

INTERVENTIONS:
Drug: Netarsudil Ophthalmic Solution 0.02% — 1 drop in each eye once daily in the evening
  Other Names: Rhopressa

SUMMARY:
To evaluate the IOP lowering efficacy of netarsudil ophthalmic solution 0.02% when used as monotherapy or when used concomitantly with other IOP-lowering agents in subjects with elevated IOP due to open angle glaucoma or ocular hypertension in a real-world clinical setting. The study is an open-label design. The patients will receive treatment for 12 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female subjects (aged 18 or older)
2. Subjects diagnosed with open-angle glaucoma or ocular hypertension, and determined by the treating physician to require additional intraocular pressure (IOP)-lowering treatment with netarsudil 0.02%.
3. Willingness to follow protocol requirements, including signed informed consent, routine follow-up schedule, completing questionnaires and completing laboratory tests

Key Exclusion Criteria:

1. Have any active ocular disease other than glaucoma or ocular hypertension that would interfere with study interpretation
2. Women of childbearing potential who are pregnant, nursing, or planning a pregnancy and not using a medically acceptable form of birth control. Male subjects with a female partner of childbearing potential must have had a prior vasectomy or agree to use an effective method of birth control during the treatment period and for 3 months after the subject has completed the study.
3. Known sensitivity or allergy to the study medication or components
4. Any systemic disease or clinical evidence of any condition which would make the subject, in the opinion of the investigator, unsuitable for the study or could potentially confound the study results
5. Concurrent participation or prior participation in any investigational drug or device study within the last 30 days prior to the Baseline Visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2018-12-27 (Actual); Primary Completion 2019-07-26 (Actual); Study Completion 2019-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Hollander, MD, MBA, Study Director — Aerie Pharmaceuticals, Inc.
Locations (22):
- United States (22):
  - Atlantis Eyecare, Huntington Beach, California
  - Harvard Eye Associates, Laguna Hills, California
  - North Bay Eye Associates, Inc, Petaluma, California
  - Shettle Eye Research Inc, Largo, Florida
  - Center For Sight, Sarasota, Florida
  - Coastal Research Associates, LLC, Roswell, Georgia
  - Wheaton Eye Clinic, Ltd, Wheaton, Illinois
  - Stiles Eyecare Excellence and Glaucoma Institute, PA, Overland Park, Kansas
  - Gaddie Eye Centers, LLC, Louisville, Kentucky
  - Glaucoma Consultants, Baltimore, Maryland
  - Tekwani Vision Center, St Louis, Missouri
  - Mark J. Weiss, M.D., Inc., Tulsa, Oklahoma
  - Scott & Christie and Associates, PC, Cranberry Township, Pennsylvania
  - Valley Eye Professionals, LLC, Huntingdon Valley, Pennsylvania
  - Carolina Cataract & Laser Center, Ladson, South Carolina
  - Total Eye Care, PA, Memphis, Tennessee
  - VRF Eye Specialty Group, Memphis, Tennessee
  - Advancing Vision Research, Nashville, Tennessee
  - Keystone Research, Austin, Texas
  - Cataract & Glaucoma Center, El Paso, Texas
  - Houston Eye Associates, Houston, Texas
  - The Eye Centers of Racine and Kenosha, Racine, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zaman F, Gieser SC, Schwartz GF, Swan C, Williams JM. A multicenter, open-label study of netarsudil for the reduction of elevated intraocular pressure in patients with open-angle glaucoma or ocular hypertension in a real-world setting. Curr Med Res Opin. 2021 Jun;37(6):1011-1020. doi: 10.1080/03007995.2021.1901222. Epub 2021 Mar 27. PMID 33733980

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 261 subjects were enrolled across 22 investigational sites and 260 treated.
Pre-assignment Details: The enrolled population includes all subjects who signed ICF. One subject enrolled but withdrew consent before study drug dispensed; thus, post-baseline treatment is unavailable. Participant Flow data represents ITT population. Clarification of enrolled (n= 261) vs treated (n=260) subjects is provided in Recruitment & Pre-assignment sections.
Groups:
- Netarsudil Ophthalmic Solution 0.02% Monotherapy: Netarsudil Ophthalmic Solution 0.02% Monotherapy: 1 drop in each eye once daily in the evening.
- Netarsudil Ophthalmic Solution 0.02% Concomitant Therapy: Netarsudil Ophthalmic Solution 0.02% - Used Concomitantly With Other IOP Lowering Agents (2-5 total agents used). 1 drop in each eye once daily in the evening.
Period: Overall Study
Arm/Group | Netarsudil Ophthalmic Solution 0.02% Monotherapy | Netarsudil Ophthalmic Solution 0.02% Concomitant Therapy
Started | 99 | 161
Completed | 81 | 138
Not Completed | 18 | 23
Not completed — Adverse Event | 13 | 17
Not completed — Lack of Efficacy | 2 | 0
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Intolerance to Conjunctival Hyperemia | 1 | 0
Not completed — IOP Too High | 1 | 1
Not completed — IOP Too High, Nerve/Visual Field Changes | 0 | 1
Not completed — Visit Out of Window | 0 | 1
Not completed — Medication Non-Compliance | 0 | 1

BASELINE CHARACTERISTICS:
Population: Modified intent to treat (mITT) population included all subjects who received at least 1 dose of study medication and had at least 1 follow-up visit with a completed IOP measurement.
Groups:
- Netarsudil Ophthalmic Solution 0.02% Monotherapy: Netarsudil Ophthalmic Solution 0.02% Monotherapy - 1 drop in each eye once daily in the evening.
- Total: Total of all reporting groups
Arm/Group | Netarsudil Ophthalmic Solution 0.02% Monotherapy | Netarsudil Ophthalmic Solution 0.02% Concomitant Therapy | Total
Number analyzed (Participants) | 91 | 151 | 242
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.2 (11.85) | 67.2 (10.53) | 67.2 (11.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 91 | 148
  Male | 34 | 60 | 94
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 8 | 19
  Not Hispanic or Latino | 80 | 143 | 223
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 45 | 58
  White | 77 | 102 | 179
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure (IOP)
Description: Percent Change from Baseline IOP at Week 12, as measured by Goldmann applanation tonometry.
  Prostaglandin analog (PGA). Fixed dose combination (FDC).
Time Frame: 12 weeks
Population: Modified Intent-to-Treat (mITT) population included all subjects who received at least 1 dose of study medication and had at least 1 follow-up visit with a completed IOP measurement.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Netarsudil Ophth Sol 0.02% Monotherapy - Tx Naïve At Baseline: During study Netarsudil Ophthalmic Solution 0.02% Monotherapy - Treatment naïve at baseline visit. 1 drop in each eye once daily in the evening.
- Netarsudil Ophth Sol 0.02% Monotherapy - Replaced 1 Agent: During study Netarsudil Ophthalmic Solution 0.02% Monotherapy - Replaced 1 agent at baseline visit (majority were PGA replacements). 1 drop in each eye once daily in the evening.
- Netarsudil Ophth Sol 0.02% Monotherapy - Replaced 2 Agents: During study Netarsudil Ophthalmic Solution 0.02% Monotherapy - Replaced 2 agents at baseline visit (including PGA and FDC replacements). 1 drop in each eye once daily in the evening.
- Netarsudil Ophth Sol 0.02% Concomitant Therapy: During study Netarsudil Ophthalmic Solution 0.02% - Used concomitantly with other IOP lowering agents (2-5 total agents used). 1 drop in each eye once daily in the evening.
Arm/Group | Netarsudil Ophth Sol 0.02% Monotherapy - Tx Naïve At Baseline | Netarsudil Ophth Sol 0.02% Monotherapy - Replaced 1 Agent | Netarsudil Ophth Sol 0.02% Monotherapy - Replaced 2 Agents | Netarsudil Ophth Sol 0.02% Concomitant Therapy
Number analyzed (Participants) | 24 | 61 | 6 | 151
percent change | -16.9 (16.35) | -2.3 (16.23) | 0.2 (8.81) | -17.0 (16.81)
Statistical Analysis 1: Comparison: Netarsudil Ophth Sol 0.02% Monotherapy - Tx Naïve At Baseline vs Netarsudil Ophth Sol 0.02% Monotherapy - Replaced 1 Agent vs Netarsudil Ophth Sol 0.02% Monotherapy - Replaced 2 Agents vs Netarsudil Ophth Sol 0.02% Concomitant Therapy; Cohorts assessed versus baseline treatment; Test type: Other — Descriptive statistics included the number of subjects/eyes(n), mean, SD, median, minimum, and maximum for continuous variables, and frequency and percentages for categorical variables; All efficacy data were summarized at each timepoint using appropriate descriptive statistics for the overall populations as well as separately for monotherapy and concomitant therapy groups

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during the course of the 12-week treatment period.
Description: The safety population included all subjects who received at least 1 dose of study medication.
Groups:
- Netarsudil Ophthalmic Solution 0.02% Monotherapy: Netarsudil Ophthalmic Solution 0.02% Monotherapy. 1 drop in each eye once daily in the evening.
Arm/Group | Netarsudil Ophthalmic Solution 0.02% Monotherapy | Netarsudil Ophthalmic Solution 0.02% Concomitant Therapy
All-Cause Mortality (participants affected / at risk) | 0/99 | 0/161
Serious Adverse Events (participants affected / at risk) | 2/99 | 1/161
Other Adverse Events (participants affected / at risk) | 43/99 | 58/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Netarsudil Ophthalmic Solution 0.02% Monotherapy (N=99) | Netarsudil Ophthalmic Solution 0.02% Concomitant Therapy (N=161)
Cellulitis Lower Left Extremity (Infections and infestations) | 0 (0) | 1 (1)
Malignant Melanoma of Eyelid (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Netarsudil Ophthalmic Solution 0.02% Monotherapy (N=99) | Netarsudil Ophthalmic Solution 0.02% Concomitant Therapy (N=161)
Conjunctival Hyperemia (Eye disorders) | 22 (22) | 32 (32)
Vision Blurred (Eye disorders) | 9 (9) | 10 (10)
Conjunctival Hemorrage (Eye disorders) | 6 (6) | 8 (8)
Instillation Site Pain (Eye disorders) | 6 (6) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-12-18): https://cdn.clinicaltrials.gov/large-docs/88/NCT03808688/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-15): https://cdn.clinicaltrials.gov/large-docs/88/NCT03808688/SAP_001.pdf